CLINICAL TRIAL: NCT05175378
Title: Adherence to Mediterranean Diet and Cardiovascular Health in Multiple Sclerosis Female Patients: a Case Control Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iaso Maternity Hospital, Athens, Greece (Other)
Collaborators: Harokopio University (Other); G.Gennimatas General Hospital (Other)
Responsible Party: Principal Investigator, Panos Papandreou, Dr., Iaso Maternity Hospital, Athens, Greece
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: #E31052019
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Multiple Sclerosis
Keywords: relapsing-remitting multiple sclerosis; Mediterranean diet; cardiovascular health
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Intervention Model Description: Randomized, case control study
Who Masked: Participant, Investigator
Masking Description: * All patients were randomly assigned to either the control or the intervention group, using single randomization. An independent researcher applied a computerized sequence to generate the randomization list. Next, the principal investigator who was responsible for the completion of each participant's form recorded the patient trial number in a sealed envelope. Maintenance of the blind-to-treatment allocation was performed in order to avoid bias. Treatment data were exposed to the analyst only after assessing outcomes. During the 3-month intervention, dietitians performed regular phone interviews on a 15-day basis to assist nutritional and lifestyle consultation in both groups.
  * All patients were instructed to keep (a) weekly food diaries (2 weekdays and 1 weekend day) and (b) 24-hour dietary records, which all were assessed remotely via emails and unexpected phone calls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Active Comparator): In the intervention group, MS women received a personalized daily eating plan (specific meals, recipes, food portions) together with nutritional consultation on the Meditteranean dietary pattern, as well as physical activity guidelines. All essential aspects of the dietary plan e.g. daily energy expenditure, classification of physical activity based on the concept of metabolic equivalent (MET), caloric adjustment according to nutritional status, and macronutrient distribution were calculated by a Clinical Decision Support System (CDSS). Body mass index (BMI) was also calculated, as the ratio of reported weight (kg) to the square of height (m2). Co-existed health issues, such as constipation or esophageal reflux, were taken into consideration. All MS patients acquired personal login passwords that allowed them to get access to their personal CDSS account and track their progress in regards to body weight, physical activity, and healthy food choices consumption.
  Interventions: Other: Lifestyle intervention
- Control arm (Sham Comparator): Patients of the control group received general dietary advice and physical activity recommendation that was in accordance with the "National Dietary Guidelines for Greek adults"
  Interventions: Other: Lifestyle intervention

INTERVENTIONS:
Other: Lifestyle intervention — We investigated the potential cardiovascular health effects of the Mediterranean dietary pattern on adult women with relapsing-remitting multiple sclerosis, in regards to body weight, body composition, cardiovascular blood biomarkers (fasting glucose, lipids, C-reactive protein), as well as depression and anxiety levels.

SUMMARY:
Multiple sclerosis (MS) is a chronic immune-mediated neurodegenerative disease that affects the central nervous system (CNS). The exact pathophysiology of MS remains unclear; it is suggested that the inflammatory state persists under a genetic-energetic-environmental complex causing a variety of clinical symptoms depending on the neuroanatomical location of MS lesions. The age of MS onset ranges between 20 and 40 years. MS is usually initiated as a relapsing-remitting disease, which may last several years to decades affecting females twice as often as males. Dietary factors may have an important impact on MS. Data from human and animal studies indicate that saturated fatty acids (SFA), the major fat type of animal foods in the "Western" diet, increase MS susceptibility. The Mediterranean dietary (MedDiet) pattern is hypothesized to be beneficial to MS patients protecting against the development cardiovascular diseases. However, little is known about the cardiovascular effects of the MedDiet on MS patients. Consequently, the aim of the present randomized, case control study was to investigate the effects of MedDiet on cardiovascular factors in women with relapsing-remitting MS after a 3-month intervention period.

DETAILED DESCRIPTION:
* Adult women with MS, who were outpatients of Iaso Hospital (Athens, Greece), were enrolled in the present study. Detailed information was provided using a leaflet, in which aims and methodology were described before recruitment. All participants fulfilled informed consent and kept a signed copy. Before the start of the trial, the Ethics Committee of Iaso Hospital (Athens, Greece) assessed and approved the protocol of the study (Approval Code #E31052019). The study was performed according to principles of the Helsinki Declaration (1964) and terms of Good Clinical Practice.
* The study took place during the winter season. All patients were recruited at the first week of December 2020 and the intervention lasted 3 months.
* Study design: 3-month randomized, single center case control study; maintenance of the blind-to-treatment allocation was performed in order to avoid bias; in the intervention group, MS women received a personalized daily eating plan generated by a Clinical Decision Support System (CDSS) together with nutritional consultation on the Meditteranean dietary pattern, as well as physical activity guidelines; patients of the control group received general dietary advice and physical activity recommendation that was in accordance with the "National Dietary Guidelines for Greek adults";
* Screening: medical history; nutritional history (food frequency questionnaire, MedDietScore, 24-hr recalls); anthropometrics; depression and anxiety (Hospital Anxiety and Depression Scale); blood biomarkers (glucose, lipids, C-reactive protein).

ELIGIBILITY:
Inclusion Criteria: adult women (≥ 18 years) with relapsing-remitting MS diagnosis; patients should follow a standardized immunomodulatory therapy or other disease-modifying therapy for at least 6 months; the patient should be able to walk without aid or work a full day in a position of average difficulty, as indicated by scores of Expanded Disability Status Scale (EDSS) < 4.5; patients with at least one lesion on brain MRI and/or at least one relapse in the past two years.

Exclusion Criteria: women with concomitant illness (e.g. malignancy, infections, malabsorption, heart-, liver- or renal failure); patients who changed treatment during or ≤ 6 months before the start or the trial; psychiatric conditions, alcoholism, drug addiction; using vitamin or mineral supplements during or ≤ 6 months prior to screening; following a vegan diet ≤ 5 years prior to screening or using weight loss medications; pregnant or lactating women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
MedDietScore | 3 months
  The MedDietScore questionnaire estimated the degree of adherence to MD at the start of the study and at 3 months. Scoring ranges from "0" to "55" and higher scores signify greater MD adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- Iaso Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No